CLINICAL TRIAL: NCT06659198
Title: Assessing the Perioperative Outcomes of Minimally Invasive Posterior Approach Versus Direct Anterior Approach Total Hip Arthroplasty: a Prospective Comparative Randomized Study on Blood and Pain Management.
Brief Title: Assessing the Perioperative Outcomes of Minimally Invasive Posterior Approach Versus Direct Anterior Approach Total Hip Arthroplasty.
Acronym: PTACONF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Collaborators: Istituto Clinico San Siro (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PTACONF
Record Dates: First submitted 2024-10-18; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Total Hip Replacement Surgery
Keywords: total hip replacement; minimally invasive posterolateral approach; direct anterior approach; blood management
MeSH Terms: interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- minimally invasive posterior approach (Experimental): minimally invasive posterior approach total hip replacement
  Interventions: Procedure: total hip replacement
- direct anterior approach (Experimental): direct anterior approach total hip replacement
  Interventions: Procedure: total hip replacement

INTERVENTIONS:
Procedure: total hip replacement — minimally-invasive hip replacement

SUMMARY:
The aim of the present study is to compare the early post-operative outcomes of minimally invasive posterolateral approach (Mis-PLA) Vs. direct anterior approach (DAA) in the treatment of primary hip osteoarthritis, with regards to blood loss and postoperative pain.

Fifty patients treated with THA from 2022 to 2023 are randomly assigned to either receive Mis-PLA or DAA THA. Visual Analog Scale (VAS) is used to assess pain and recorder ad hospital admission and on postoperative days 1 and 3. Intraoperative and postoperative blood loss and blood transfusion rate are recorded, as well as operation time and length of stay (LOS).

DETAILED DESCRIPTION:
Total hip arthroplasty (THA) is considered a reliable surgical strategy for the treatment of end-stage hip osteoarthritis, although it is associated with postoperative complications, such as perioperative pain and blood loss sometimes leading to blood transfusions. Recently, the concept of enhanced recovery surgery in minimally invasive joint replacement surgery is gaining popularity, as opposed to traditional approaches, which possess disadvantages such as a higher risk of dislocation, longer hospital stays and rehabilitation periods, and increased soft tissue injuries.

The minimally invasive posterolateral approach (Mis-PLA) with preserved piriformis muscle was found to minimize the amount of time needed for functional recovery, preserve prosthesis stability, reduce postoperative pain, and cause less injury and perioperative blood loss when compared to the standard procedure. It has a number of benefits, such as a very simple procedure, a clearly visible surgical field, less damage to soft tissues, and better abductor muscle preservation.

Similarly, the direct anterior approach (DAA) offers several advantages like a lower risk of dislocation, quick recovery, and less intraoperative muscle injury, although according to some studies, it possesses a longer learning curve and it is associated with prolonged operation times and significant perioperative bleeding.

This study compares the early post-operative outcomes of Mis-PLA Vs. DAA in the treatment of primary hip osteoarthritis, with regards to blood loss and postoperative pain.

Fifty patients suffering from hip osteoarthritis treated with THA from 2022 to 2023 constitute the study sample size. Patients are subdivided into two groups and randomly assigned to either receive Mis-PLA or DAA THA.

Patients should be included if they comply with the following criteria: unilateral primary or secondary end-stage hip osteoarthritis candidate to THA, body mass index<30 kg/m2, American Society of Anesthesiologists (ASA) grade <3, absence of liver disease, coagulative pathology. Exclusion criteria are as follows: ASA grade ≥ 3, history of bleeding or thrombotic disorder, history of liver or renal disease, anticoagulant or antiplatelet therapy, refusal to participate in the study.

Patients eligible for randomization are randomly assigned to either group with a random number table randomization. Patients are followed-up up to 45 days after surgery to evaluate the occurrence of perioperative complications. This study was approved by the ethics committee of IRCCS San Raffaele Hospital, Milan, Italy, on 18/7/19 (approval number 2016005).

Patient demographics and anthropometric characteristics (age, sex, operated side, BMI) are recorded. The length of stay is calculated from admission until discharge. Peripheral blood samples are collected preoperatively and on postoperative days 1 and 3. Visual Analog Scale (VAS) is used to assess pain and recorder ad hospital admission and on postoperative days 1 and 3. Total blood loss and blood transfusion rate are also recorded, as well as operation time. Blood transfusion is administered at a haemoglobin threshold of 8 g/dl in patients without comorbidities, and a threshold of 10 g/dl in patients with pre-existing cardiac pathology, according to international guidelines.

Surgical procedure of the Mis-PLA:

Following spinal anesthesia, patients are placed in lateral decubitus on the unaffected side. A short longitudinal oblique incision over the posterior aspect of the greater trochanter is performed. The sciatic nerve and gluteus medius are then shielded, the subcutaneous tissue and the underlying fascia of the tensor fasciae lata are severed, and a retractor is applied to lift the piriformis muscle upwards. After detachment of obturator internus, gemelli and quadratus, joint capsulotomy is performed. The hip is dislocated and osteotomy of the neck performed in the usual fashion. The acetabular margin is cleaned to expose the bony landmarks. Uncemented prostheses are then placed in the acetabular cup and into the femural shaft.

Surgical procedure of the DAA:

Patients are positioned supine on the table, after spinal anaesthesia is induced. A longitudinal slightly oblique incision is made on the anterior-lateral aspect of the thigh, starting 2 cm distal and lateral to the ASIS. After subcutaneous fat and fascia dissection, the interval between the tensor muscle and the rectus femoris is identified. Lateral femoral circumflex vessels are ligated and anterior hip capsule incised. After neck osteotomy and femoral head extraction, reaming, and cup placement is performed, followed by femoral preparation and stem insertion. The fascia over the tensor is stitched with sutures. Skin closure is performed and a sterile dressing is applied through a drainage previously positioned.

Peri-operative and rehabilitation protocol:

Both groups receive the same perioperative management. Antibiotics (2g of cefazolin sodium) administered intravenously before surgery. The patients are given a pre-operative dose of 15 mg/ kg tranexamic before surgery, and 15 mg/kg of the medication into the joint cavity after skin closure. Following surgery, a cold pack is placed over the surgical incision and compressive socks used. To prevent venous thromboembolism, low molecular weight heparin (LMWH) is administered subcutaneously 8 h after surgery, and prolonged up to 30 days after operation.

Postoperative oral celecoxib or other non-steroidal anti-inflammatory edication as needed are part of the postoperative pain regimen.

Patients are instructed to start early isometric quadriceps exercises and ankle pump exercises, walking with partial weight bearing with the use of crutches from the first day after surgery.

Statistical analysis Data are analyzed using Graphpad Prism v8.0 (Prism Software, La Jolla, CA, USA). Data distribution analysis is performed using the Shapiro-Wilk test. The t-test is used to analyze normally distributed data from the two groups; non parametric Mann-Withney test is used in case of non-normal distribution of data. Categorical variable are expressed as absolute and relative frequency and have been compared using Fisher's exact test. Differences are deemed statistically significant with p value < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* clinical and instrumented diagnosis of unilateral primary or secondary end-stage hip osteoarthritis candidate to total hip arthroplasty
* patients with body mass index<30 kg/m2,
* absence of liver disease, coagulative pathology

Exclusion Criteria:

* patients with history of bleeding or thrombotic disorder,
* patients with history of liver or renal disease
* patients with anticoagulant or antiplatelet therapy
* refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Number of participants requiring blood tranfusions | preop to 3 days postop
  Number (percentage) of participants requiring blood tranfusions

SECONDARY OUTCOMES:
Visual analog scale (VAS) score for each patient | preop to 3 days postop
  Visual analog scale (VAS) rates pain severity froma a scale of 0 (no Pain) to 10 (worst pain possible)

OTHER OUTCOMES:
Number and type of intra- and post-operative complications | Up to 30 days after surgery
  Number and type of intra- and post-operative complications

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Galeazzi, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided